CLINICAL TRIAL: NCT01549171
Title: Pilot Study to Examine Iloprost Can Enhance Human Assisted Reproductive Technology Pregnancy Outcomes.
Brief Title: Enhanced Assisted Reproductive Technology Pregnancy Rate by Prostacyclin Analog (Iloprost)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fertility Specialists of Houston (Other)
Collaborators: Origio A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: OGAFSH-01
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Pregnancy
Keywords: Human ART; Prostacyclin; Iloprost; Pregnancy
MeSH Terms: interventions — Iloprost; Saline Solution

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Iloprost: This is the study group with 1 uM Iloprost.
  Interventions: Drug: Iloprost
- Control: This is the control group with vehicle (normal saline) only.
  Interventions: Other: normal saline

INTERVENTIONS:
Drug: Iloprost — supplement in culture medium during culture in the lab. The concentration is 1 uM.
  Other Names: Ilomedin
  Groups: Iloprost
Other: normal saline — Supplement with vehicle only no Iloprost.
  Groups: Control

SUMMARY:
Human fallopian tube secretes high concentration of prostacyclin. Fallopian tube is the site for early embryo development. The effect of prostacyclin on human early embryo development is waiting to be clarified. The study hypothesis is prostacyclin can enhance early embryo development.

DETAILED DESCRIPTION:
Huang et al, found that human fallopian tube expresses prostacyclin synthetase and cyclooxygenase. These enzyme systems synthesize abundant prostacyclin (PGI2). In the fallopian tube PGI2 causes smooth muscle relaxation, possibly facilitating tubal transport of gametes and embryos. Huang et al reported that addition of the PGI2 analogue Iloprost to embryo culture media significantly enhanced mouse embryo development to the blastocyst and complete hatched stages. The implantation and live birth rates of Iloprost cultured embryos were significantly better than non-Iloprost embryos in the mouse model. The mean weights of fetal mice were not significant different from control group. There was no teratogenic effect observed.

In a previously presented study, the investigators cultured donated frozen human zygotes in culture media with and without the addition of Iloprost. The Iloprost treated embryos showed significantly better growth rate and morphology, as determined by the size, and grading of the trophectoderm and inner cell mass.

Iloprost is FDA approved for the treatment of pulmonary hypertension. It has a significantly longer half-life than native PGI2. Iloprost is a class C pregnancy drug and has not been associated with teratogenic effects. This study intends to expand the usage of Iloprost to culture embryos.

ELIGIBILITY:
Inclusion Criteria:

* ART case

Exclusion Criteria:

* age < 40
* no pre-implantation genetic diagnosis procedure

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: ART cases with age < 40 and without pre-implantation genetic diagnosis
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-11 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Presence of embryo sac in uterus under ultrasound | 5 weeks after embryo transfer
  The competency of embryo is determined by its ability to implant into endometirum.

SECONDARY OUTCOMES:
The delivery outcome is the secondary outcome measured. | 10 months after embryo transfer
  The live birth and the weight and length of baby is examined.

CONTACTS AND LOCATIONS:
Overall Officials: George M Grunert, M.D., Principal Investigator — Obstetrical & Gynecological Associates
Locations (1):
- Fertility Specialists of Houston, Houston, Texas, United States

REFERENCES:
- [Background] Battenfeld R, Schuh W, Schobel C. Studies on reproductive toxicity of iloprost in rats, rabbits and monkeys. Toxicol Lett. 1995 Aug;78(3):223-34. doi: 10.1016/0378-4274(95)03323-d. PMID 7542807
- [Background] Grunert GM, Dunn RC, Valdes CT, Schenk LM, Mangal RK, Wun WSA: Prostacyclin agonist (Iloprost) enhances human embryo development. Fertility and Sterility 84:S237, 2005
- [Background] Huang JC, Arbab F, Tumbusch KJ, Goldsby JS, Matijevic-Aleksic N, Wu KK. Human fallopian tubes express prostacyclin (PGI) synthase and cyclooxygenases and synthesize abundant PGI. J Clin Endocrinol Metab. 2002 Sep;87(9):4361-8. doi: 10.1210/jc.2002-020199. PMID 12213900
- [Background] Huang JC, Wun WS, Goldsby JS, Matijevic-Aleksic N, Wu KK. Cyclooxygenase-2-derived endogenous prostacyclin enhances mouse embryo hatching. Hum Reprod. 2004 Dec;19(12):2900-6. doi: 10.1093/humrep/deh524. Epub 2004 Oct 15. PMID 15489241
- [Background] Huang JC, Goldsby JS, Wun WS. Prostacyclin enhances the implantation and live birth potentials of mouse embryos. Hum Reprod. 2004 Aug;19(8):1856-60. doi: 10.1093/humrep/deh352. Epub 2004 Jun 17. PMID 15205402